CLINICAL TRIAL: NCT05918055
Title: A Phase I/II Trial of Eltanexor (KPT-8602) With Inqovi (Decitabine-Cedazuridine) in High-Risk Myelodysplastic Syndromes
Brief Title: Eltanexor (KPT-8602) With Inqovi (Decitabine-Cedazuridine) in High-Risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug company withdrew support.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Najla El Jurdi, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001541; 001541-C
Record Dates: First submitted 2023-06-23; First posted 2023-06-26 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Acute Myeloid Leukemia; hypomethylating agents; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Eltanexor; decitabine and cedazuridine drug combination; Decitabine; cedazuridine; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I- Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes (Experimental): Inqovi for 5 days, followed by escalating doses of Eltanexor (KPT-8602)
  Interventions: Drug: KPT-8602; Drug: Inqovi; Procedure: Bone marrow aspirate; Procedure: Bone marrow biopsy; Diagnostic Test: ECG
- Phase II- Dose expansion for High-Risk Myelodysplastic Syndromes (Experimental): Inqovi for 5 days, followed by recommended phase 2 dose (RP2D)/Phase II dose of Eltanexor (KPT-8602)
  Interventions: Drug: KPT-8602; Drug: Inqovi; Procedure: Bone marrow aspirate; Procedure: Bone marrow biopsy; Diagnostic Test: ECG

INTERVENTIONS:
Drug: KPT-8602 — 5-10 mg by mouth (PO) daily for 10-14 days based on dose level
  Other Names: Eltanexor
Drug: Inqovi — Inqovi will be administered via oral route once daily on Days 1-5 of each treatment cycle, according to guidelines outlined in the Food and Drug Administration (FDA) product label.
  Other Names: Decitabine; Cedazuridine
Procedure: Bone marrow aspirate — Screening (if necessary), baseline (30 days prior to treatment start), and Cycle 1, Day 28 (phase I only).
  Other Names: BM aspirate
Procedure: Bone marrow biopsy — Screening (if necessary), baseline (30 days prior to treatment start), and Cycle 1, Day 28 (phase I only).
  Other Names: BM biopsy
Diagnostic Test: ECG — Screening and baseline. Cycle 1, Day 1 and Cycle 1, Day 15 (2 hours post dose that day +/- 20 minutes).
  Other Names: Electrocardiogram

SUMMARY:
Background:

Myelodysplastic syndromes (MDS) are diseases that affect the bone marrow. They can inhibit the blood formation process and reduce blood cell counts. High-risk MDS can lead to leukemia. People with high-risk MDS have a low survival rate. Better treatments are needed.

Objective:

To test a study drug Eltanexor (KPT-8602), combined with another drug (Inqovi), in people with MDS.

Eligibility:

Adults aged 18 years and older with high-risk MDS that did not respond to treatment.

Design:

Participants will be screened. They will have a physical exam. They will have blood and urine tests and tests of their heart function. They may have a bone marrow biopsy: Their hip will be numbed; then a needle will be inserted to draw out a sample of soft tissue from inside the bone. They will answer questions about their quality of life. Genetic tests may be performed.

KPT-8602 and Inqovi are both tablets taken by mouth. Participants will take these drugs at home on a 28-day cycle. They will take Inqovi once a day on days 1 to 5. They will take KPT-8602 on a schedule assigned by the researcher. Participants will be given a drug diary to record each dose.

Participants will visit the clinic for an exam at least once in each cycle. Some tests, including the bone marrow biopsy, may be repeated.

Participants will continue treatment for at least 6 cycles. If their disease improves, they may continue taking the drugs after 6 cycles.

Participants will have follow-up visits at the clinic for about 8 years.

DETAILED DESCRIPTION:
Background:

* The myelodysplastic syndromes (MDS) are a group of clonal bone marrow neoplasms characterized by ineffective hematopoiesis, cytopenia, and high risk of transformation to acute myeloid leukemia (AML).
* The median survival of patients with newly diagnosed higher-risk MDS (HR-MDS) according to the Revised International Prognostic Scoring System (IPSS-R) is 1.5 years.
* Hypomethylating agents (HMAs), such as azacitidine and decitabine, are the standard of care therapy for HR-MDS. However, less than half of patients respond to HMAs, and even the best responses are transient and non-curative.
* The only curative treatment for patients with MDS is allogeneic hematopoietic stem cell transplantation (HSCT); however, only a small portion are eligible for transplant.
* More effective therapies are needed for patients with HR-MDS.
* A promising approach for improving HMA efficacy in the treatment of MDS is by exploiting therapeutic synergism in combinatorial approaches.
* Inqovi (decitabine-cedazuridine) is an oral formulation of decitabine plus cytidine deaminase inhibitor that was recently Food and Drug Administration (FDA)-approved for MDS, based on a similar safety and efficacy profile to decitabine for injection.
* KPT-8602 (eltanexor) is an orally available, second-generation selective inhibitor of nuclear export (SINE) that covalently binds to exportin 1 (XPO1).
* XPO1 is a protein that mediates the nuclear export of molecules from the nucleus to the cytoplasm of the cell. Among affected molecules are tumor suppressor genes, messenger ribonucleic acid (mRNAs) encoding oncogenes (including cellular myelocytomatosis oncogene (c-MYC), and newly assembled ribosomal subunits.
* By interfering with c-MYC translation, KPT-8602 may diminish rebound methylation after decitabine cessation and improve treatment responses in patients with MDS.
* Preliminary reports from a Phase 1/2 trial of KPT-8602 monotherapy in patients with higher-risk MDS who have failed HMAs show anti-tumor activity and an acceptable toxicity profile.
* Sequential addition of KPT-8602 to Inqovi may improve treatment responses in patients with MDS by acting synergistically to inhibit further DNA methylation.

Objective:

* Phase I: To determine the recommended phase 2 dose (RP2D) of KPT-8602 in combination with Inqovi in adult participants with higher-risk MDS
* Phase II: To determine overall response rate (ORR) of KPT-8602 in combination with Inqovi in adult participants with higher- risk MDS

Eligibility:

* Participants must have histologically or cytologically confirmed MDS according to 2016 World Health Organization (WHO) criteria, and for both Phase I and II:
* have HR-MDS (Revised International Prognostic Scoring System (IPSS-R) > 3.5) with inadequate response to hypomethylating agent (HMA) therapy (received >= 4 cycles of the standard dose (35 mg decitabine and 100 mg cedazuridine) without prior dose-reductions, with failure to achieve at least a PR or experienced disease progression prior to completing 4 cycles)
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2 (KPS >= 60)

Design:

* Participants with HR-MDS will be enrolled in both Phase I and II.
* Participants will be treated with Inqovi at a fixed dose of 1 tablet (35 mg decitabine and 100 mg cedazuridine) daily on Days 1-5 of each 28-day cycle, followed by KPT-8602 at escalating doses (Phase I) or the RP2D (Phase II).
* In Phase I, KPT-8602 will be dose-escalated following a standard 3+3 design, with a starting dose level of 10 mg for 10 days (staggered) within a cycle. If tolerated, the dose will be escalated to 14 days per cycle, or dose de-escalated to 5 mg at 14 or 10 days.
* This study will be done at the National Institutes of Health (NIH) Center with an enrollment of up to 80 planned participants.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Participants must have histologically or cytologically confirmed Myelodysplastic Syndromes (MDS) by the Laboratory of Pathology, NCI- according to 2016 World Health Organization (WHO) criteria AND:

   -Cohort 1 (Phase 1) & 2 (Phase 2): have high-risk Myelodysplastic Syndromes (HR-MDS) Revised International Prognostic Scoring System (IPSS-R > 3.5) with inadequate response to hypomethylating agent (HMA) therapy [(received >= 4 cycles of the standard dose (35 mg decitabine and 100 mg cedazuridine) without prior dose reductions, with failure to achieve at least a partial remission (PR) or experienced disease progression prior to completing 4 cycles)
2. Age >=18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status <= 2 (Karnofsky >= 60%,)
4. Participants must have adequate organ and marrow function as defined below:

   -total bilirubin <= 1.5 X institutional upper limit of normal

   OR

   <= 3 X institutional upper limit of normal in participants with Gilbert's syndrome (except for participants with increased bilirubin levels attributed to intramedullary hemolysis, which will be allowable)

   -Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine transaminase (ALT) serum glutamic pyruvic transaminase (SGPT) <= 3 X institutional upper limit of normal

   OR

   <= 5 X institutional upper limit of normal if related to MDS-specific cause
   * creatinine clearance (by Cockcroft-Gault) >= 60 mL/min/1.73m^2
   * corrected QT interval using the Fridericia formula (QTc(F) <= 470 ms
5. Individuals of child-bearing potential (IOCBP) must have a negative serum test at screening. IOCBP is defined as the following:

   * Has not undergone a hysterectomy, tubal ligation, or bilateral oophorectomy
   * Has not been naturally postmenopausal for at least 24 consecutive months (i.e.,has had menses at any time in the preceding 24 consecutive months).
6. Individuals of childbearing potential (IOCBP) as well as those able to father a child with an individual able to become pregnant potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) unless they have had a prior vasectomy, hysterectomy, or bilateral oophorectomy, prior to study entry, for the duration of study participation, and for at least 6 months after last dose of HMA.
7. Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 30 days after the last administration of study drug
8. Any prior therapy must have been completed >4 weeks or, if known, >= 5 half-lives of the prior agent (whichever is shorter) prior to treatment (with a minimum of 1 week between prior therapy and study treatment). Note: This does not apply to prior HMA therapy if that therapy is Inqovi.
9. Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants with platelet transfusion-refractory thrombocytopenia, with inability to keep platelet threshold above 10K/mcL with transfusions or those with ongoing or uncontrolled hemorrhagic complications.
2. Participants with clinically significant neutropenia, defined as absolute neutrophil count (ANC) <100 cells/mcL with frequent hospitalizations for infection (average > 1 hospitalization per month in the past 6 months).
3. Participants on treatment with a myeloid growth factor (e.g., granulocyte colony-stimulating factor (G-CSF) within 14 days prior to initiation of study treatment.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to HMAs, or other agents used in study.
5. Uncontrolled intercurrent illness evaluated by history, physical exam, and chemistries or situations that would limit compliance with study requirements, interpretation of results or that could increase risk to the participant
6. Participants with the following cardiac conditions: symptomatic congestive heart failure, unstable angina pectoris, or uncontrolled cardiac arrhythmia as assessed by electrocardiogram (ECG).
7. Pregnancy (confirmed with Beta-human chorionic gonadatropin (HCG) serum or urine pregnancy test performed in individuals of childbearing potential at screening)
8. Presence of any other malignancy (except basal and squamous cell carcinoma of the skin, or stable chronic cancers on hormone or targeted therapy) for which participant received systemic anticancer treatment (except maintenance therapy) within 24 months prior to treatment.
9. Participants with active/uncontrolled Hepatitis B
10. Participants with active/uncontrolled Hepatitis C
11. Participants with active/uncontrolled human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
12. Participants currently taking contraindicated medications for HIV, Hepatitis B, or Hepatitis C disease control

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be shared. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Data from this study may be requested by contacting the principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001541-C.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All (#3) participants enrolled in this study are counted. 1/3 participants were deemed ineligible after consent was signed to participate in the study. Baseline data for this participant was collected and reported. All participants that started Dose Level 1 were de-escalated to Dose Level -1
Groups:
- Phase I - Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes: Inqovi for 5 days, followed by escalating doses of Eltanexor (KPT-8602)
  KPT-8602: 5-10 mg by mouth (PO) daily for 10-14 days based on dose level
  Inqovi: Inqovi will be administered via oral route once daily on Days 1-5 of each treatment cycle, according to guidelines outlined in the Food and Drug Administration (FDA) product label.
- Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes: Inqovi for 5 days, followed by recommended phase 2 dose (RP2D)/Phase II dose of Eltanexor (KPT-8602)
  KPT-8602: 5-10 mg by mouth (PO) daily for 10-14 days based on dose level
  Inqovi: Inqovi will be administered via oral route once daily on Days 1-5 of each treatment cycle, according to guidelines outlined in the Food and Drug Administration (FDA) product label.
- Participant Enrolled But Not Treated: Participant was enrolled but not treated.
Period: Phase I - Dose Level 1
Arm/Group | Phase I - Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes | Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes | Participant Enrolled But Not Treated
Started | 2 | 0 | 1
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 1
Period: Phase I - Dose Level -1
Arm/Group | Phase I - Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes | Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes | Participant Enrolled But Not Treated
Started | 2 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Phase II
Arm/Group | Phase I - Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes | Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes | Participant Enrolled But Not Treated
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 participants were started in Dose Level 1 and were deescalated to Dose level - 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes | Participant Enrolled But Not Treated | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (16.26) | 81 (0) | 56.67 (24.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity - Hispanic or Latino | 2 | 0 | 2
  Ethnicity - Not Hispanic or Latino | 0 | 1 | 1
  Ethnicity - Unknown or Not Reported | 0 | 0 | 0
  Race - American Indian or Alaska Native | 0 | 0 | 0
  Race - Asian | 0 | 0 | 0
  Race -Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race - Black or African American | 0 | 0 | 0
  Race - White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Race - Unknown or Not Reported | 1 | 0 | 1
  Race - Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D) of Eltanexor (KPT-8602) in Combination With Inqovi (Decitabine-Cedazuridine) in Adult Participants With Higher-Myelodysplastic Syndromes (MDS)
Description: If no DLTs are observed at the highest planned dose level for evaluation (dose level 2), dose escalation will stop, and this will be considered the recommended phase 2 dose (RP2D) of Eltanexor (KPT-8602). A DLT is defined as a treatment-related toxicity based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: From day 1 of study drug through 28 days after the first dose
Population: 2/3 participants were analyzed because the 2 participants that started in Dose Level 1, also de-escalated and treated on Dose Level -1. And 1 participant were not treated in Dose Level 1 or Dose Level-1 because they were not eligible for the study.
Measure: Number; unit: mg
Groups:
- All Participants in Phase I: All participants in phase I who received at least 9/10 doses of Eltanexor (KPT-8602) and 4/5 doses of Ingovi (Decitabine-Cedazuridine) within the DLT period.
Arm/Group | All Participants in Phase I
Number analyzed (Participants) | 2
mg | NA — The RP2D was not found because the number of participants accrued was inadequate to establish a RP2D.

2. Primary Outcome: Phase 1: Number of Participants Who Have Grades 3 and/or 4 Dose-limiting Toxicity (DLT) at the Recommended Phase 2 Dose (RP2D)
Description: Participants enrolled in phase I will have the grades and types of toxicity reported at each dose level to determine the RP2D. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event. Toxicity was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Time Frame: First 28 days of study treatment
Population: 2/3 participants were analyzed because one participant was enrolled but not treated.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I:Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1: Participants with confirmed Myelodysplastic Syndromes and International Prognostic Scoring System (IPSS-R) score >3.5 (high and higher intermediate-risk).
  Dose level 1: Ingovi (Decitabine-Cedazuridine), 1 tablet orally once daily on Days 1-5. Eltanexor (KPT-8602), 10 mg by mouth (PO) daily on Days 8-12 and Days 15-19.
- Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1: Participants with confirmed Myelodysplastic Syndromes and International Prognostic Scoring System (IPSS-R) score >3.5 (high and higher intermediate-risk).
  Dose level -1: Ingovi (Decitabine-Cedazuridine), 1 tablet orally once daily on Days 1-4. Eltanexor (KPT-8602) 5 mg by mouth (PO) daily on Days 8-21.
Arm/Group | Phase I:Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 | Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1
Number analyzed (Participants) | 2 | 2
Participants
  Grade 3 Platelet Count Decreased | 1 | 0
  Grade 4 Platelet Count Decreased | 1 | 0
  Grade 4 Neutrophil Count Decreased | 1 | 0

3. Primary Outcome: Phase 2: Overall Response Rate (ORR) of Eltanexor (KPT-8602) in Combination With Inqovi (Decitabine-Cedazuridine) Reported With a 95% Confidence Interval in Adult Participants With Higher-Myelodysplastic Syndromes (MDS)
Description: Participants evaluated in phase II will have the fraction with clinical responses reported, with a 95% confidence interval. ORR is defined as Complete Remission (CR)+Partial Remission (PR)+marrow (mCR) with hematologic improvement (HI) per each cohort and assessed by the 2006 International Working Group Response Criteria with Modified Definitions for Hematologic Improvement by the 2018 International Working Group Response Criteria. Complete Remission (CR) is bone marrow: ≤5% myeloblasts with normal maturation of all cell lines. Partial Remission (PR) is all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pretreatment but still >5%; and cellularity and morphology not relevant. Marrow Complete Remission is bone marrow: ≤5% myeloblasts and decrease by ≥50% over pretreatment.
Time Frame: Each cycle (bloods), cycle 2 and 6 during treatment and every 3-6 months (bloods and bone marrow)
Population: This outcome was not done because no participants accrued on phase 2.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes: Inqovi for 5 days, followed by recommended phase 2 dose (RP2D)/Phase II dose of Eltanexor (KPT-8602) KPT-8602: 5-10 mg by mouth (PO) daily for 10-14 days based on dose level Inqovi: Inqovi will be administered via oral route once daily on Days 1-5 of each treatment cycle, according to guidelines outlined in the Food and Drug Administration (FDA) product label.
  Bone marrow aspirate: Screening (if necessary), baseline (30 days prior to treatment start), and Cycle 1, Day 28 (phase I only).
  Bone marrow biopsy: Screening (if necessary), baseline (30 days prior to treatment start), and Cycle 1, Day 28 (phase I only).
  ECG: Screening and baseline. Cycle 1, Day 1 and Cycle 1, Day 15 (2 hours post dose that day +/- 20 minutes).
Arm/Group | Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1: AUC Under the Concentration Time Curve (AUC 0-48h) of Eltanexor (KPT-8602) in Combination With Inqovi (Decitabine-Cedazuridine) in Participants With Myelodysplastic Syndromes (MDS)
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: 1, 2, 3, 4, 8, 24 and 48 hours after the product administration on days 8 and 21 of cycle one
Population: Data was not analyzed and reported because samples collected are insufficient to complete analysis. Since 2 participants were accrued to study this drug has been removed from analysis by the drug company. No further studies are becoming completed, and the samples will not be analyzed in the future.
Measure: Mean (Standard Deviation); unit: Mg*h/mL
Arm/Group | Phase I:Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 | Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase 1: Half-life of Eltanexor (KPT-8602) in Combination With Inqovi (Decitabine-Cedazuridine) in Participants With Myelodysplastic Syndromes (MDS)
Description: The half-life of Eltanexor (KPT-8602) will be evaluated in participants, by dose level when given in combination with Inqovi. Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: 1, 2, 3, 4, 8, 24 and 48 hours after the product administration on days 8 and 21 of cycle one
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1: Participants with confirmed Myelodysplastic Syndromes and International Prognostic Scoring System (IPSS-R) score >3.5 (high and higher intermediate-risk).
  Dose level 1: Ingovi (Decitabine-Cedazuridine), 1 tablet orally once daily on Days 1-5. Eltanexor (KPT-8602), 10 mg by mouth (PO) daily on Days 8-12 and Days 15-19.
Arm/Group | Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 | Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 1: Calculating Steady State (Css) Concentration of Eltanexor (KPT-8602) When Given in Combination With Inqovi (Decitabine-Cedazuridine)
Description: Steady state concentration, measured by the Eltanexor (KPT-8602) blood concentration will be evaluated in participants, by dose level when given in combination with Inqovi (Decitabine-Cedazuridine). Steady state is defined as consistent drug concentration in the body.
Time Frame: 1, 2, 3, 4, 8, 24 and 48 hours after the product administration on days 8 and 21 of cycle one
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Phase I:Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 | Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 2: Number of Grades 1, 2, 3, 4, and/or 5 Toxicity of Eltanexor (KPT-8602) and Inqovi (Decitabine-Cedazuridine) at Each Dose Level in Participants With Myelodysplastic Syndromes (MDS)
Description: The grades and types of toxicity noted for the agent at each dose level will be reported. Toxicity was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: At least weekly through cycle 3 and then at the start and every cycle after that
Population: This outcome was not done because no participants accrued on phase 2.
Measure: Number; unit: toxicity
Arm/Group | Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 2: Number of Serious Adverse Events Leading to Discontinuation, Death, and Laboratory Abnormalities
Description: A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Serious adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Time Frame: At least weekly through cycle 3 and then at the start and every cycle after that
Population: This outcome was not done because no participants accrued on phase 2.
Measure: Number; unit: adverse events
Arm/Group | Phase II - Dose expansion for High-Risk Myelodysplastic Syndromes
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Phase 1: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From the first study intervention through 30 days after the study agent (s) was/were administered, an average of 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I:Dose escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 | Phase I:Dose escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1 | Participant Enrolled But Not Treated
Number analyzed (Participants) | 2 | 2 | 1
Participants | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed an average of 8.5 months. Adverse Events were monitored/assessed from the first study intervention through 30 days after the study agent (s) was/were administered, an average of 8.5 months.
Description: Dosages on Dose Level -1 and Dose Level 1 were administered to participants during treatment. Start date is Start Date of 1st Course, cutoff date is Date Off Treatment. Adverse Events (AEs) can happen before treatment, during treatment and after treatment. Most of the AEs happened during the treatment in this study. There are only 4 Adverse Events for one participant which happened after Date Off Treatment (Outside Courses).
Groups:
- Outside Courses: One participant experienced 4 adverse events that occurred after Date Off Treatment (Outside Courses).
Arm/Group | Phase I:Dose Escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 | Phase I:Dose Escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1 | Participant Enrolled But Not Treated | Outside Courses
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I:Dose Escalation of Eltanexor (KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level 1 (N=2) | Phase I:Dose Escalation of Eltanexor(KPT-8602) for High-Risk Myelodysplastic Syndromes-Dose Level -1 (N=2) | Participant Enrolled But Not Treated (N=1) | Outside Courses (N=1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (10) | 2 (13) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (4) | 1 (2) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Stomach discomfort after taking Deferasirox. (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify: Port occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (4) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (6) | 1 (7) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify: Hepatic steatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — : Vitamin D mild deficiency 14 ng/ml (still above 10 ng/ml).
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify: Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (13) | 2 (7) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (6) | 1 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — : Burning sensation on suprapubic area during micturition
Renal and urinary disorders - Other, specify: Burning sensation when urinating (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Nocturia (1-2 urinations per night) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Polyuria, polydipsia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (10) | 2 (23) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT05918055/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT05918055/ICF_001.pdf